CLINICAL TRIAL: NCT06413147
Title: Long-term Procedural and Device Related Complications of PFO Closure
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, yinchunlin, Xuanwu Hospital, Capital Medical University, Xuanwu Hospital, Beijing
Other Study IDs: yinchunlin_PFO safety
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: PFO closure — Surgery of PFO closure

SUMMARY:
We aimed to explore: (1）long-term complications of PFO closure; (2) antiplate or anticoagulation use after PFO closure.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent PFO closure

Exclusion Criteria:

* Unable to complete or adhere to the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent PFO closure and willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke, Hemorrhagic stroke or transient ischemic attack | 1 month, 6 months, 1 year, 3 years, 5 years

SECONDARY OUTCOMES:
atrial fibrillation | 1 month, 6 months, 1 year, 3 years, 5 years
Hemorrhage related to the use of antithrombotic drugs | 1 month, 6 months, 1 year, 3 years, 5 years
residual leaks | 1 month, 6 months, 1 year, 3 years, 5 years
death | 1 month, 6 months, 1 year, 3 years, 5 years
open-heart surgery | 1 month, 6 months, 1 year, 3 years, 5 years
Other severe events related to PFO closure | 1 month, 6 months, 1 year, 3 years, 5 years

IPD SHARING:
Plan to Share IPD: No